CLINICAL TRIAL: NCT03776253
Title: Conquer Fear SUPPORT: A Psychosocial Intervention in Patients With Advanced Cancer
Brief Title: Conquer Fear SUPPORT Intervention in Supporting Patients With Stage III-IV Lung or Gynecologic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18305; NCI-2018-02405 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18305 (Other: City of Hope Medical Center)
Record Dates: First submitted 2018-10-31; First posted 2018-12-14 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Advanced Lung Carcinoma; Malignant Female Reproductive System Neoplasm; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (CFS) (Experimental): Patients attend CFS psychosocial intervention consisting of 7 nurse-led sessions (session 1 in-person and sessions 2-7 via video conferencing) over 45 minutes each for 8 weeks. Patients also complete home practice assignments comprising attention training technique and mindfulness practice after each session.
  Patients complete self-report questionnaires at baseline (T1), 8 weeks (T2) and 12 weeks (T3).
  Interventions: Behavioral: Psychosocial Care Conquer Fear Support intervention (psychoeducation, attention training, worry management, and detached mindfulness components); Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Psychosocial Care Conquer Fear Support intervention (psychoeducation, attention training, worry management, and detached mindfulness components) — Attend CFS
  Other Names: Conquer Fear Support
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial will pilot a psychosocial intervention called Conquer Fear Support (CFS) in patients with stage III-IV lung or gynecologic cancer who are experiencing fear of cancer progression. The intervention is adapted from a novel program called "Conquer Fear" which was developed by researchers in Australia. CFS may help in reducing worries, fears, and uncertainty in patients with advanced lung or gynecological cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the feasibility and acceptability of the CFS intervention in patients with advanced lung and gynecologic (GYN) cancer (stages III or IV) who have clinically significant levels of fear of cancer progression (FOP) or cancer-related distress.

SECONDARY OBJECTIVES:

I. Assess preliminary effects of the intervention on FOP, cancer-specific distress, anxiety, depression, overall symptom distress, metacognitions, and mindfulness.

OUTLINE:

Patients attend CFS psychosocial intervention consisting of 7 nurse-led sessions (session 1 in-person and sessions 2-7 via video conferencing) over 45 minutes each for 8 weeks. Patients also complete home practice assignments comprising attention training technique and mindfulness practice sessions after each session.

After completion of study intervention, patients are followed up at week 12.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gynecologic (GYN) and lung cancer will be recruited
* Stage III or IV disease
* At least 3 months from initial diagnosis
* Receiving disease-focused treatment or active surveillance mode
* A score of ≥ 34 on the Fear of Progression Questionnaire-Short Form (SF) or ≥ 24 on the Impact of Event Scale-Revised
* All subjects must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Current severe depression or psychosis; significant cognitive impairment
* Patients enrolled in hospice care or who opt to receive no further disease-focused treatment
* Patients who are currently receiving ongoing psychiatric treatment
* Non-English speaking

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Conquer Fear SUPPORT (CFS) intervention is assessed by tracking enrollment rate. | Up to 9 months
  Evaluate the enrollment (recruitment) rate over the study period. Feasibility will be deemed acceptable if at least 25 eligible participants are accrued within 9 months.
Feasibility of the Conquer Fear SUPPORT (CFS) intervention is assessed by tracking attrition. | Up to week 12
  Evaluate attrition (drop-out rate) over time for enrolled participants. Feasibility will be deemed acceptable if the percentage of patients who drop-out does not exceed 20% by week 8 of the intervention and 50% by week 12 of the intervention.
Feasibility of the Conquer Fear SUPPORT (CFS) intervention is assessed by tracking attendance. | Up to week 12
  Evaluate the percentage of sessions attended. Feasibility will be deemed acceptable if participants attend an average of 5 of the 7 scheduled sessions.

SECONDARY OUTCOMES:
Fear of progression (FOP) assessed using Fear of Progression Questionnaire-Short Form (SF) | Up to week 12
  Fear of progression will be assessed using Fear of Progression Questionnaire-Short Form (FOP-Q-SF) at baseline (T1), 8 weeks (T2), and 12 weeks (T3).
  FOP-Q-SF consists of 12 items scored on a 5-point Likert scale (1=never to 5=very often); scores range from 12-60 with higher levels indicating greater FOP. Researchers have used a cut-off of 34 and above to indicate dysfunctional FOP.
Cancer-specific distress assessed using the Impact of Event Scale-Revised (IES-R) | Up to week 12
  Cancer-specific distress will be assessed using the Impact of Event Scale-Revised (IES-R) at baseline (T1), 8 weeks (T2), and 12 weeks (T3). IES-R is a 22-item scale consisting of 3 subscales a) Intrusion; b) Avoidance; and c) Hyperarousal. Items are scored on a 0-4 response format. Subscale scores are calculated by taking the mean of the subscale responses. Total scores range from 0-88. A score of 24 or greater indicates clinical levels of distress.
Anxiety assessed using the PROMIS-Anxiety 8a | Up to week 12
  Anxiety will be assessed using the PROMIS-Anxiety 8a at baseline (T1), 8 weeks (T2), and 12 weeks (T3). PROMIS-Anxiety measures fear, dread, worry, hyperarousal, and related somatic symptoms. The short-form consists of 8 items that are scored on a 0-5 response format. The raw score is calculated by summing the values of the response to each question (range 8-40). Scores are standardized such that the scale produces continuous T scores with a mean of 50 and a SD of 10, higher scores reflect higher distress. PROMIS T score thresholds for anxiety are: ˂ 55 normal; 55-64 mild; 65-74 moderate; ≥75 severe.
Depression assessed using the Patient Health Questionnaire (PHQ-9) | Up to week 12
  Depression will be assessed using the Patient Health Questionnaire (PHQ-9) at baseline (T1), 8 weeks (T2), and 12 weeks (T3). The PHQ-9 includes the two major symptom domains: affective and somatic symptoms. It is rated from a 0 (not at all) to 3 (nearly every day) scale. Items are summed and a score of 10 or greater is considered clinically significant symptoms of depression. Scores of 0-4, 5-9, 10-14, and ≥15 represent minimal, mild, moderate, and severe levels of symptom burden.
Overall symptom distress assessed using the Memorial Symptom Assessment Scale (MSAS) | Up to week 12
  Overall symptom distress will be assessed using the Memorial Symptom Assessment Scale (MSAS) at baseline (T1), 8 weeks (T2), and 12 weeks (T3). The MSAS assesses 32 common symptoms experienced by cancer patients. A modified version of the MSAS will be used to evaluate the occurrence, severity, and distress of symptoms. Symptom severity is rated on a 4 point Likert scale (1=slight) to 4=very much). Distress is rated on a 0-4 Likert scale ranging from not at all (0) to very much (4). The physical symptom subscale is the average of the severity and distress associated with 12 physical symptoms. The psychological symptom subscale is the average of the severity and distress associated with 6 psychological symptoms. The total MSAS score (TMSAS) is the average of the symptom scores of all 32 symptoms; higher scores indicate greater symptom severity and distress.
Metacognitions (MCQ-30) assessed using the Metacognitions Questionnaire | Up to week 12
  Metacognitions (MCQ-30) will be assessed using the Metacognitions Questionnaire at baseline (T1), 8 weeks (T2), and 12 weeks (T3). The MCQ-30 is a 30-item questionnaire that assesses beliefs about worry. It consists of 5 subscales: Positive beliefs about worry; Negative beliefs about worry, Cognitive confidence; Need to control thoughts; and Cognitive self-consciousness. For each subscale, items are scored 1-4 and subscale scores range from 6-24. Total scores range from 30 to 120; higher scores indicate more dysfunctional metacognitions.
Mindfulness assessed using the Five Facet Mindfulness Questionnaire (FFMQ-15) | Up to week 12
  Mindfulness will be assessed using the Five Facet Mindfulness Questionnaire (FFMQ-15) at baseline (T1), 8 weeks (T2), and 12 weeks (T3). The FFMQ-15 assesses five facets of mindfulness: observing, describing, acting with awareness, non-reactivity, and non-judging of inner experience. Items are rated on a 5-point Likert scale ranging from 1 (never or rarely true) to 5 (very often or always true). 3 items comprise each subscale and subscale scores range from 3-15. Higher scores indicate greater engagement with mindfulness skills.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Reb, NP, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States